CLINICAL TRIAL: NCT01215786
Title: Safety and Pharmacodynamics Study of AGN-207281 Ophthalmic Solutions Compared With Timolol Ophthalmic Solution or Placebo in Patients With Ocular Hypertension or Primary Open-Angle Glaucoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 207281-004
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Results first posted 2012-01-16 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AGN-207281 ophthalmic solution (Other): AGN-207281 0.1% ophthalmic solution on Days 1-7 and AGN-207281 0.3% ophthalmic solution on Days 8-14
  Interventions: Drug: AGN-207281 ophthalmic solutions (0.1% and 0.3%); AGN-207281 vehicle ophthalmic solution (placebo)
- Timolol ophthalmic solution 0.5% (Active Comparator): timolol ophthalmic solution 0.5%
  Interventions: Drug: timolol ophthalmic solution 0.5%
- Placebo (Placebo Comparator): AGN-207281 vehicle ophthalmic solution (Placebo)
  Interventions: Drug: AGN-207281 vehicle ophthalmic solution (Placebo)

INTERVENTIONS:
Drug: AGN-207281 ophthalmic solutions (0.1% and 0.3%); AGN-207281 vehicle ophthalmic solution (placebo) — One drop of AGN-207281 ophthalmic solutions (0.1% on Days 1-7 and 0.3% on Days 8-14) instilled to both eyes in the morning followed by one drop of AGN-207281 vehicle ophthalmic solution (placebo) instilled to both eyes in the evening for 13 days.
  Arms: AGN-207281 ophthalmic solution
Drug: timolol ophthalmic solution 0.5% — One drop of timolol ophthalmic solution 0.5% instilled to both eyes, in the morning for 14 days, and in the evening for 13 days
  Arms: Timolol ophthalmic solution 0.5%
Drug: AGN-207281 vehicle ophthalmic solution (Placebo) — One drop of AGN-207281 vehicle ophthalmic solution instilled to both eyes, in the morning for 14 days and in the evening for 13 days.
  Arms: Placebo

SUMMARY:
This is an exploratory study that will evaluate the safety and pharmacodynamics of up to 3 doses of AGN-207281 based on an ongoing review of data during the study period compared with timolol ophthalmic solution or placebo in patients with ocular hypertension or primary open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension or primary open-angle glaucoma in each eye
* Requires IOP-lowering therapy in both eyes
* Visual acuity score of 20/100 or better in each eye

Exclusion Criteria:

* Experienced significant weight change (over 10 pounds) within 60 days
* History of alcohol or drug addiction
* History of migraines or frequent headaches
* Anticipated wearing of contact lenses during the study
* Required chronic use of ocular medications during study
* Eye surgery within 6 months
* Use of systemic beta blockers (eg, atenolol, propranolol) within 2 months
* Use of oral, intramuscular, intravenous corticosteroids within 21 days
* Use of ophthalmic corticosteroids within 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients in the AGN-207281 ophthalmic solution arm received AGN-207281 ophthalmic solution 0.1% on Days 1 to 7 and AGN-207281 ophthalmic solution 0.3% on Days 8 to 14.
Period: Overall Study
Arm/Group | AGN-207281 Ophthalmic Solution | Timolol Ophthalmic Solution 0.5% | Placebo
Started | 21 | 19 | 10
Completed | 21 | 19 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-207281 Ophthalmic Solution | Timolol Ophthalmic Solution 0.5% | Placebo | Total
Number analyzed (Participants) | 21 | 19 | 10 | 50
Age, Customized [Number; unit: participants]
  <45 years | 0 | 0 | 1 | 1
  Between 45 and 65 years | 7 | 7 | 2 | 16
  >65 years | 14 | 12 | 7 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 7 | 28
  Male | 8 | 11 | 3 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Worse Eye Intraocular Pressure (IOP) at Day 14
Description: Change from baseline in worse eye IOP at day 14. Worse eye IOP refers to the eye with the worse (highest) baseline IOP (a measurement of the fluid pressure inside the eye). A negative number change from baseline indicates a reduction in IOP (improvement).
Time Frame: Baseline, Day 14
Population: Safety population, which consisted of all patients who started the study and received treatment.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mm Hg)
Arm/Group | AGN-207281 Ophthalmic Solution | Timolol Ophthalmic Solution 0.5% | Placebo
Number analyzed (Participants) | 21 | 19 | 10
Millimeters of mercury (mm Hg)
  Baseline, Hour 0 | 25.98 (2.581) | 26.58 (2.673) | 26.45 (2.661)
  Baseline, Hour 2 | 25.93 (3.207) | 26.61 (3.125) | 26.30 (2.781)
  Baseline, Hour 8 | 24.69 (2.610) | 24.82 (2.578) | 25.25 (2.889)
  Change from Baseline at Day 14, Hour 0 | -4.17 (2.825) | -6.16 (3.189) | -1.10 (2.039)
  Change from Baseline at Day 14, Hour 2 | -4.38 (3.244) | -6.08 (2.955) | -1.75 (2.690)
  Change from Baseline at Day 14, Hour 8 | -4.02 (2.826) | -4.00 (3.000) | -1.70 (1.814)

2. Secondary Outcome: Mean Concentration of AGN-207281 in Plasma at Day 7
Description: Mean concentration of AGN-207281 in plasma at day 7. Plasma is the liquid component of the blood in which the blood cells are suspended. On day 7, the plasma sample collected 15 minutes post-morning dose from each patient receiving AGN-207281 was analyzed to determine the average drug concentration levels of AGN-207281.
Time Frame: Day 7
Population: The analysis population included all patients that started the study and were treated with AGN-207281.
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | AGN-207281 Ophthalmic Solution | Timolol Ophthalmic Solution 0.5% | Placebo
Number analyzed (Participants) | 21 | 0 | 0
Picograms per milliliter (pg/mL) | 177 (113) |  |

3. Secondary Outcome: Mean Concentration of AGN-207281 in Plasma at Day 14
Description: Mean concentration of AGN-207281 in plasma at day 14. Plasma is the liquid component of the blood in which the blood cells are suspended. On day 14, the plasma sample collected 15 minutes post-morning dose from each patient receiving AGN-207281 was analyzed to determine the average drug concentration levels of AGN-207281.
Time Frame: Day 14
Population: The analysis population included all patients that started the study and were treated with AGN-207281.
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | AGN-207281 Ophthalmic Solution | Timolol Ophthalmic Solution 0.5% | Placebo
Number analyzed (Participants) | 21 | 0 | 0
Picograms per milliliter (pg/mL) | 540 (263) |  |

ADVERSE EVENTS:
Arm/Group | AGN-207281 Ophthalmic Solution | Timolol Ophthalmic Solution 0.5% | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/10
Other Adverse Events (participants affected / at risk) | 9/21 | 19/19 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-207281 Ophthalmic Solution (N=21) | Timolol Ophthalmic Solution 0.5% (N=19) | Placebo (N=10)
Eye irritation (Eye disorders) | 7 | 8 | 0
Eye pain (Eye disorders) | 1 | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 2 | 0
Punctate keratitis (Eye disorders) | 0 | 4 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo